CLINICAL TRIAL: NCT03315702
Title: the Change of R-spondin Proteins Plasma Concentration Level Caused by Mechanical Ventilation and Its Effect on Mechanical Ventilation Induced Lung Injury
Brief Title: Effect of Mechanical Ventilation on Plasma Concentration Level of R-spondin Proteins
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-17-015
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Results first posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2017-10

CONDITIONS: Acute Lung Injury
Keywords: R-spondin proteins, mechanical ventilation, lung injury
MeSH Terms: conditions — Acute Lung Injury; Lung Injury | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood samples from patients undergo elective surgery with general anesthesia and mechanical ventilation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- control／mechanical ventilation: venous blood samples collected from patients twice，relatively before mechanical ventilation and 3rd hour after mechanical ventilation
  Interventions: Other: mechanical ventilation

INTERVENTIONS:
Other: mechanical ventilation — mechanical ventilation protocol: tidal volume 6-8 ml/kg, positive end-expiratory pressure 5 cm H2O, oxygen concentration 40%; respiratory rate 10-15/min, inspiratory/expiratory ratio 1:1.5.

SUMMARY:
As novel agonists of Wnt/β-catenin signaling pathway, R-spondin proteins constitute a class of ligands, including R-spondin 1/2/3/4, functioning through their receptors leucine-rich repeat-containing G-protein coupled receptor (LGR)4/5/6 to enhance Wnt/β-catenin activity. Since Wnt signaling plays pivotal roles in the regulation of many life processes involved in embryogenesis and adulthood, R-spondin proteins also take part in cell proliferation, differentiation and morphogenesis.For example, in the formation of respiratory system，R-spondin 2 is required for normal laryngeal-tracheal and lung morphogenesis，and the lack of R-spondin 1 expression results in the absence of duct side-branching development and subsequent alveolar formation. In addition, R-spondins show protective effect in tissue injury and diseases. R-spondin 1 and R-spondin 3 have been reported to prevent chemotherapy- or radiotherapy-induced mucous membrane lesion. R-spondin 1 attenuates oral mucositis contributed by radiotherapy in mouse models and R-spondin 3 potentiates intestinal regeneration elicited via gastrointestinal toxic effect of chemoradiotherapy treatment. However, whether R-spondin proteins exert salient influence on acute lung injury especially induced by mechanical ventilation is deficient. Therefore, this study aims to ascertain the implication of R-spondin proteins in the pathology of mechanical ventilation induced lung injury through detecting human plasma concentration change of R-spondin 1/2/3/4 after mechanical ventilation and interference effects in mouse model, which is helpful for prevention and treatment of ventilation induced lung injury.

DETAILED DESCRIPTION:
Mechanical ventilation is a critical intervention for patients with acute respiratory failure. However, lung overdistension induced by mechanical ventilation also causes pulmonary endothelial dysfunction. The injurious effect of mechanical stretch on pulmonary endothelium has been implicated in the development of ventilator-induced lung injury, which is characterized by pulmonary inflammation and particularly increased vascular permeability. In addition, the investigators and others have previously shown that mechanical stretch increases cultured lung endothelial monolayer permeability in vitro and promotes lung vascular permeability in mice Thus, elucidating the mechanisms underlying the mechanical stretch-induced lung endothelial barrier dysfunction may provide a novel clinical therapeutic target against ventilator-induced lung injury.

As novel agonists of Wnt/β-catenin signaling pathway, R-spondin proteins constitute a class of ligands, including R-spondin 1/2/3/4, functioning through their receptors leucine-rich repeat-containing G-protein coupled receptor (LGR)4/5/6 to enhance Wnt/β-catenin activity. Since Wnt signaling plays pivotal roles in the regulation of many life processes involved in embryogenesis and adulthood, R-spondin proteins also take part in cell proliferation, differentiation and morphogenesis. For example, in the formation of respiratory system，R-spondin 2 is required for normal laryngeal-tracheal and lung morphogenesis，and the lack of R-spondin 1 expression results in the absence of duct side-branching development and subsequent alveolar formation. In addition, R-spondins show protective effect in tissue injury and diseases. R-spondin 1 and R-spondin 3 have been reported to prevent chemotherapy- or radiotherapy-induced mucous membrane lesion. R-spondin 1 attenuates oral mucositis contributed by radiotherapy in mouse models and R-spondin 3 potentiates intestinal regeneration elicited via gastrointestinal toxic effect of chemoradiotherapy treatment. However, whether R-spondin proteins exert salient influence on acute lung injury especially induced by mechanical ventilation is deficient. Therefore, this study aims to ascertain the implication of R-spondin proteins in the pathology of mechanical ventilation induced lung injury through detecting human plasma concentration change of R-spondin 1/2/3/4 after mechanical ventilation and interference effects in mouse model, which is helpful for prevention and treatment of ventilation induced lung injury.

ELIGIBILITY:
Inclusion Criteria:

* undergo elective surgery with mechanical ventilation lasting for > 3 hours; classified as physical status I to III according to the American Society of Anesthesiologists Physical Status Classification System; Written informed consent is approved.

Exclusion Criteria:

* chronic lung disease; recent lung infection; recent anaesthetics or mechanical ventilation treatment; hemodilution with massive fluid supply during surgery; children；women during pregnancy or lactation; being involved in other clinical subjects

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients undergo elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lai Jiang, chief doctor, Study Chair — Xinhua Hospital affiliated to Medicine school,Shanghai Jiaotong University
Locations (1):
- Department of Anesthesia, Shanghai Xinhua hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control／Mechanical Ventilation
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Control／Mechanical Ventilation
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 52
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Concentration of R-spondin 1
Description: The venous blood samples were collected twice for each patient that the first time was around the onset of the mechanical ventilation and the second was 3rd hour after the onset of the mechanical ventilation, which were named as sample A and sample B relatively. Then, plasmids were separated by centrifugation and detected for R-spondin1 concentration. And the outcome was calculated by subtracting the R-spondin1 plasmid concentration of sample A from the R-spondin1 plasmid concentration of sample B, which was the change in plasma concentration of R-spondin1.
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Control／Mechanical Ventilation: Venous blood samples collected from patients twice before mechanical ventilation and 3rd hour after
  mechanical ventilation: mechanical ventilation protocol: tidal volume 6-8 ml/kg, positive end-expiratory pressure 5 cmH2O, oxygen concentration 40%; respiratory rate 10-15/min, inspiratory/expiratory ratio 1:1.5.
Arm/Group | Control／Mechanical Ventilation
Number analyzed (Participants) | 52
pg/ml | 1407.4080 (1350.7859)

2. Primary Outcome: Change in Plasma Concentration of R-spondin 2
Description: The venous blood samples were collected twice for each patient that the first time was around the onset of the mechanical ventilation and the second was 3rd hour after the onset of the mechanical ventilation, which were named as sample A and sample B relatively. Then, plasmids were separated by centrifugation and detected for R-spondin2 concentration. And the outcome was calculated by subtracting the R-spondin2 plasmid concentration of sample A from the R-spondin2 plasmid concentration of sample B, which was the change in plasma concentration of R-spondin2.
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control／Mechanical Ventilation
Number analyzed (Participants) | 52
pg/ml | -2.1830 (35.3601)

3. Primary Outcome: Change in Plasma Concentration of R-spondin3
Description: The venous blood samples were collected twice for each patient that the first time was around the onset of the mechanical ventilation and the second was 3rd hour after the onset of the mechanical ventilation, which were named as sample A and sample B relatively. Then, plasmids were separated by centrifugation and detected for R-spondin3 concentration. And the outcome was calculated by subtracting the R-spondin3 plasmid concentration of sample A from the R-spondin3 plasmid concentration of sample B, which was the change in plasma concentration of R-spondin3.
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control／Mechanical Ventilation
Number analyzed (Participants) | 52
pg/ml | -2.8956 (30.2781)

4. Primary Outcome: Change in Plasma Concentration of R-spondin4
Description: The venous blood samples were collected twice for each patient that the first time was around the onset of the mechanical ventilation and the second was 3rd hour after the onset of the mechanical ventilation, which were named as sample A and sample B relatively. Then, plasmids were separated by centrifugation and detected for R-spondin4 concentration. And the outcome was calculated by subtracting the R-spondin4 plasmid concentration of sample A from the R-spondin4 plasmid concentration of sample B, which was the change in plasma concentration of R-spondin4.
Time Frame: 3 hours
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control／Mechanical Ventilation
Number analyzed (Participants) | 52
pg/ml | -269.8598 (1230.6612)

ADVERSE EVENTS:
Time Frame: 3 hours Explanation: The venous blood samples were collected twice for each patient that the first time was around the onset of the mechanical ventilation and the second was 3rd hour after the onset of the mechanical ventilation.
Description: Samplings of 1 ml blood were performed twice per patient from peripheral venous catheter: the first just before endotracheal intubation and the second 3rd hour after that. Systematic monitoring, including electrocardiograph monitoring, brain electricity guardianship, blood gas，blood pressure, etc., was performed during surgery process. Patients responded normally with stable postoperative consciousness. No death, serious or other adverse events occurred during this process in surgical room.
Groups:
- Control／Mechanical Ventilation: Venous blood samples were collected twice for each patient，relatively before onset of mechanical ventilation and 3rd hour after mechanical ventilation.
Arm/Group | Control／Mechanical Ventilation
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control／Mechanical Ventilation (N=52)
0 (General disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03315702/Prot_SAP_002.pdf
  • Informed Consent Form (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03315702/ICF_003.pdf